CLINICAL TRIAL: NCT06266364
Title: Targeted Plasticity Therapy for the Treatment of Post-Traumatic Stress Disorder
Brief Title: Targeted Plasticity Therapy for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Dr. Seth Hays, Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-24-22; HT94252310818 (Other Grant/Funding Number: CDMRP); 175181 (Other: The University of Texas Health Science Center at San Antonio)
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: PTSD, Post Traumatic Stress Disorder
Keywords: PTSD, Post-Traumatic Stress Disorder; VNS, Vagus Nerve Stimulation; TPT, Targeted Plasticity Therapy; ReStore System; PE, Prolonged Exposure Therapy; Trauma and Stressor Related Disorders; Mental Disorders; Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Combat Disorders; Trauma and Stressor Related Disorders; Mental Disorders; Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of active stimulation vs. sham stimulation for 12 sessions post randomization, followed by up to 12 sessions of open label active stimulation for all participants
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All are blinded in the RCT (Randomized Controlled Trial) phase. However, sites will need to have an unblinded programmer who is only programming the device and not collecting outcomes data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Immediate VNS Group (Active Comparator): The participants in this arm will be implanted with the device and will receive active VNS stimulations in phase 1 as well as phase 2 of the study.
  Interventions: Device: Active VNS stimulation
- Delayed VNS Group (Sham Comparator): The participants in this arm will be implanted with the device but will receive sham VNS stimulations in phase 1 of the study and active VNS in phase 2 of the study.
  Interventions: Device: Sham VNS stimulation

INTERVENTIONS:
Device: Active VNS stimulation — The subjects in this group will be implanted with the ReStore device and receive active Vagus nerve stimulation (VNS) in phase 1
  Arms: Immediate VNS Group
Device: Sham VNS stimulation — The subjects in this group will be implanted with the ReStore device and receive sham Vagus nerve stimulation (VNS) in phase 1
  Arms: Delayed VNS Group

SUMMARY:
Objectives of this study are to provide continued safety assessment for the ReStore system, and to gain further estimates of the effect size of Vagus Nerve Stimulation (VNS) therapy with Prolonged Exposure Therapy (PE) compared to PE with placebo (sham) stimulation in participants with posttraumatic stress disorder (PTSD)

DETAILED DESCRIPTION:
A prospective, multi-center, randomized, controlled, blinded trial of participants implanted with the ReStore Device for VNS Therapy.

In double-blinded Phase 1, after implantation, participants will be randomized to either active VNS stimulation or sham VNS stimulation, accompanying PE therapy twice weekly for 7 weeks (12 in-office sessions, Phase 1). The therapist and the participant will be blinded of the group assignment.

Following completion of Phase 1, all participants undergo two mid-therapy assessments and then advance to the open-label Phase 2.

In open-label Phase 2, all participants will receive up to an additional 12 sessions of PE therapy paired with active VNS stimulation, regardless of their prior assignment in Phase 1.

Post-therapy assessments will be performed 1 day, 1 month, and 6 months following the completion of the final session of PE in Phase 2.

During the in-office sessions, the therapist will use a secure smart device to deliver stimulation and record audio of the session for use during homework sessions. The smart device will automatically trigger VNS during audio homework sessions at the same times that the therapist delivered VNS during the corresponding in-office session.

Long-term assessment of safety will be performed up to four times annually for up to 2 years following the date of implant or until the device is FDA approved when possible. Safety assessment will only report on the presence of the implanted, non-active device and/or participant status during this period. Participants who experience a serious device-related adverse event will be removed from the identified risk but will continue to be monitored for 2 years or longer if the event has not resolved.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic PTSD for at least 3 months based on DSM-5 criteria
2. In the medical opinion of the Principal Investigator (PI), failed at least one adequate course of first-line PTSD treatment per American Psychological Association (APA) guidelines
3. PCL-5 score greater than 33
4. Age 22-79 years
5. Appropriate surgical candidate for VNS device implantation
6. Willing and able to comply with study protocol
7. Able to provide informed consent.

Exclusion Criteria:

1. Currently undergoing prolonged exposure therapy elsewhere
2. Concurrent participation in another interventional clinical trial
3. Prior injury to vagus nerve
4. Prior or current treatment with vagus nerve stimulation
5. Psychiatric disorders and/or cognitive impairments that would interfere with study participation, as assessed by medical evaluation
6. Moderate-High Risk of Suicide according to Columbia - Suicide Severity Rating Scale (C-SSRS) Screen Version
7. Persons with a current or past: (a) medical (psychiatric, non-psychiatric) condition, disease, disorder, injury, or disability or (b) non-medical situation or circumstance that, in the opinion of the principal investigator, study participation:

   * may pose a significant or undue risk to the person,
   * make it unlikely the person will complete all the study requirements per protocol, or
   * may adversely impact the integrity of the data or the validity of the study results
8. Persons with a neck circumference larger than 18.5 inches
9. Females of childbearing potential who are either pregnant or planning to become pregnant and who are not using, or will not agree to use medically acceptable birth control methods
10. Non-English speaking
11. As determined by the principal investigator, is under current incarceration or legal detention

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
ReStore System Safety | From surgery to up to 2 years following implantation or until the device is FDA approved, whichever comes first
  ReStore System safety by review of any adverse events

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5(fifth edition of the Diagnostic and Statistical Manual of Mental Disorders)(CAPS-5) | From baseline up to visit 33 (end of study)
  The CAPS-5 is a 30-item structured PTSD diagnostic interview that measures PTSD. Total scores range from 0-80, with higher scores indicating more severe PTSD symptoms symptoms.
PTSD Checklist for DSM-5 (PCL-5) score | From baseline up to visit 33 (end of study)
  The PCL-5 is a 20 item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Total scores range from 0-80, with higher scores indicating more severe PTSD symptoms symptoms.
PostTraumatic Cognitions Inventory (PTCI) | From baseline up to visit 33 (end of study)
  The PTCI is a 33-item instrument that assesses dysfunctional post-trauma cognitions across self, world, and self-blame to yield a total score. Total scores range from 33-231, with higher scores reflecting greater endorsement of negative posttraumatic cognitions.
Generalized Anxiety Disorder 7-item Scale (GAD-7) | From baseline up to visit 33 (end of study)
  The GAD-7 is a 7-item questionnaire that measures severity of anxiety. Total scores range from 0-21, with higher scores reflecting severe anxiety symptom levels.
Patient Health Questionnaire-9 (PHQ-9) | From baseline up to visit 33 (end of study)
  The PHQ-9 is a brief self-report measure of major depressive disorder. Total scores range from 0-27, with higher scores reflecting severe depression symptom levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Wigginton, MD, Principal Investigator — The University of Texas at Dallas; Robert Rennaker, PhD, Principal Investigator — The University of Texas at Dallas; Jasper Smits, PhD, Principal Investigator — The University of Texas at Austin; Mark Powers, PhD, Principal Investigator — Baylor Scott & White; Michael Kilgard, PhD, Principal Investigator — The University of Texas at Dallas
Locations (3):
- United States (3):
  - The University of Texas Health Austin Ambulatory Surgery Center, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Texas Biomedical Device Center, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No